CLINICAL TRIAL: NCT06743568
Title: Efficacy of Self-expandable and Balloon-expandable Valves in Patients With Ascending Aortic Dilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2486
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Aortic Stenosis; Ascending Aortic Dilatation
Keywords: Transcatheter aortic valve replacement; Balloon-expandable valve; Self-expandable valve; Aortic stenosis; Ascending aortic dilation
MeSH Terms: conditions — Aortic Valve Stenosis; Aneurysm, Ascending Aorta | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: The present study is a multi-center, open-label, two-arm randomized control trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-expandable valve group (Other): Patients who undergo transcatheter aortic valve replacement using self-expandable valves
  Interventions: Device: Transcatheter aortic valve replacement
- Balloon-expandable valve group (Other): Patients who undergo transcatheter aortic valve replacement using balloon-expandable valves
  Interventions: Device: Transcatheter aortic valve replacement

INTERVENTIONS:
Device: Transcatheter aortic valve replacement — Eligible patients will be randomized 1:1 to self-expandable valve group or balloon-expandable valve group.

SUMMARY:
This study evaluated the efficacy of self-expandable valves and balloon-expandable valves in patients with ascending aortic dilation who undergo transcatheter aortic valve replacement.

DETAILED DESCRIPTION:
Ascending aortic dilation (AAD) is a common feature in patients with aortic stenosis, especially in those with bicuspid aortic valve. According to the 2022 AHA/ACC Guideline for the Diagnosis and Management of Aortic Disease, in patients undergoing surgical aortic valve replacement who have a concomitant AAD with a maximum diameter of ≥45mm, ascending aortic replacement is reasonable when performed by experienced surgeons in a Multidisciplinary Aortic Team (Class 2a, Level B-NR). However, in patients undergoing transcatheter aortic valve replacement, the impact of ascending aortic dilation remains unclear. Therefore, we designed this multicenter prospective randomized controlled trial, aiming to assess the efficacy of self-expandable and balloon-expandable valves in patients with AAD with a maximum diameter of ≥45mm.

ELIGIBILITY:
Inclusion Criteria:

* Severe AS defined as an aortic valve area (AVA) of 1cm2 or less or an indexed AVA of 0.6 cm2/m2 or less;
* Evaluation and selection for TAVR by the multidisciplinary heart team;
* Maximum ascending aortic diameter between 45mm and 54mm on preoperative contrast-enhanced computed tomography (CT) scan
* Anatomic suitability for a transfemoral vascular access;
* Life expectancy of more than 12 months;
* Age ≥65 years.

Exclusion Criteria:

* Pure aortic regurgitation;
* History of surgical or transcatheter aortic valve replacement (valve in valve);
* History of any aortic surgery;
* Emergent surgery;
* Patients who refused to be randomized or unable to complete regular follow-up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Device success | Perioperative period
  (1) freedom from mortality; (2) successful access, delivery of the device, and retrieval of the delivery system; (3) correct positioning of a single prosthetic heart valve into the proper anatomical location; (4) freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication; (5) intended performance of the valve (mean gradient <20mmHg, peak velocity <3m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation).
30-day all-cause mortality | 30 days
  30-day all-cause mortality
30-day adverse aortic events | 30 days
  Aortic-related death, aortic dissection, or aortic rupture.

SECONDARY OUTCOMES:
1-year all-cause mortality | 1 year
  1-year all-cause mortality
1-year cardiovascular mortality | 1 year
  1-year cardiovascular mortality
1-year adverse aortic events | 1 year
  Aortic-related death, aortic dissection, or aortic rupture.
Aortic expansion rate≥3mm/year | 1 year
  The aortic expansion rate was defined by the change of AA diameter (before the procedure and at the latest follow-up) divided by the follow-up period.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - National Center for Cardiovascular Disease, China & Fuwai Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality
  - Fuwai Shenzhen Hospital, Shenzhen, Guangdong
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No